CLINICAL TRIAL: NCT02930850
Title: Spot-Check Noninvasive Hemoglobin (SpHb) Clinical Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TORR0002
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Anemia; Healthy; Pediatric ALL
MeSH Terms: conditions — Anemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test subjects (Experimental): All subjects are enrolled and receive Rad-67 Pulse oximeter sensor for measurement of hemoglobin.
  Interventions: Device: Rad-67 Pulse oximeter

INTERVENTIONS:
Device: Rad-67 Pulse oximeter — Noninvasive pulse oximeter that measures hemoglobin

SUMMARY:
The purpose study is to report on the accuracy of noninvasive hemoglobin (SpHb) as compared to hemoglobin measurements obtained from a laboratory hematology analyzer.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to report on the accuracy of the Rad-67 and DCI Mini sensor to measure SpHb as compared to hemoglobin measurements obtained from a manual HiCN analytical method and automated Beckman Coulter laboratory hematology analyzers.

ELIGIBILITY:
Inclusion Criteria:

* Age: Greater than one month
* Weight: Greater than or equal to 3kg
* The subject or the subject's legally authorized representative has given written informed consent/assent to participate in the study

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, nail polish, acrylic nails, infections, abnormalities, etc.
* Subjects deemed not suitable for the study at the discretion of the investigator
* Subjects unlikely to be able to refrain from excessive motion during data collection. Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.
* Decision-impaired adult and pediatric subjects who are unable to give consent and assent

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of hemoglobin measurement | Up to 2 hours per subject
  Accuracy willl be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Site 4, Burbank, California
  - Site 5, Burbank, California
  - Site 2, Irvine, California
  - Site 7, Lake Forest, California
  - Site 3, National City, California
  - Site 6, Torrance, California
  - Site 1, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No